CLINICAL TRIAL: NCT02299596
Title: Physsurg - a Controlled Randomized Trial on the Effect of Physical Activity in Relation to Outcome After Surgery
Brief Title: Physical Activity in Relation to Surgical Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Eva Haglind, MD, PhD, professor, Consultant Surgeon, Professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Physsurg C - the RCT
Record Dates: First submitted 2014-11-17; First posted 2014-11-24 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer; Surgery
Keywords: Colorectal neoplasm; Physical activity
MeSH Terms: conditions — Colorectal Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre and postoperative exercise (Experimental): The intervention is prehabilitation preoperatively and physical training postoperatively. During the hospital stay both groups will be treated in the same manner.
  Preoperative intervention:
  One half hour of exercise daily added to the existing daily exercise routine. The level of exercise should produce shortness of breath but the patient should be able to talk without much effort.
  Inspiratory muscle training. Thirty breaths x two twice daily. Postoperative intervention is mainly the same as preoperatively.
  Interventions: Other: Physical activity
- Control (No Intervention): Standard treatment with one exception, patients will fill in a physical activity diary

INTERVENTIONS:
Other: Physical activity — The intervention will take place both pre- and postoperatively. During the hospital stay both groups will be treated in the same manner.
  Arms: Pre and postoperative exercise

SUMMARY:
This study will compare the outcome after surgery between a group of patients that receives instructions for prehabilitation training and one group that received standard treatment.

DETAILED DESCRIPTION:
The aim of this study is to investigate whether a training program with intensified physical activity prior to and after a surgical procedure reduces the surgical-related postoperative recovery time, hospital stay, sick leave and complication rate.

A secondary aim is to investigate the effect of a training program with pre- and post- operative PA on the rate of resumption of QoL and normal physical function.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed colorectal cancer and a planned surgical procedure

Exclusion Criteria:

* HIPEC surgery, not able to give informed consent or understand the intervention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 761 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Recovery measured as physical recovery measured in questionnaire | 4-6 weeks

SECONDARY OUTCOMES:
Psychological recovery measured in a questionnaire, patient reported | 4-6 weeks and 1 year post-operatively
  Recovery
Recovery measured as time back to work | 1 year
  Recovery
Complications according to Clavien-Dindo | within 90 days
  Postoperative complications
QoL measured using SF-36 | 4-6 weeks and 1 year
  QoL according to SF-36
QoL measured using EQ-5D | 4-6 weeks and 1 year
  QoL according to EQ-5D
QoL measured using a specifically developed instrument for this study | 4-6 weeks and 1 year
  Health related QoL
Mortality | 3 and 5 years
  Long term mortality
Re-admissions | 1 year
  Hospital re-admissions
Reoperations | 1 year
  Reoperations
Total time of hospital stay | 1 year
  Length of stay
IGF-1 and IGFBP-3 | 4 weeks postopeartively
  Lab values
Postoperative pain measured with Brief Pain Inventory-Short form | 4 weeks
  Pain measured by BPI-S
Postoperative pain measured with Brief Pain Inventory-Short form | 12 months
  Pain measured by BPI-S
Health economic analysis | 4 weeks
  Health economic analysis modified according to results of primary outcome
Health economic analysis | 12 months
  Health economic analysis modified according to results of primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Eva Haglind, M.D., Ph.D., Principal Investigator — SSORG
Locations (2):
- Sweden (2):
  - Sahlgrenska University Hospital/Östra, Gothenburg
  - Dept. of Surgery, Skaraborgs Sjukhus, Skövde

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Onerup A, Li Y, Afshari K, Angenete E, de la Croix H, Ehrencrona C, Wedin A, Haglind E. Long-term results of a short-term home-based pre- and postoperative exercise intervention on physical recovery after colorectal cancer surgery (PHYSSURG-C): a randomized clinical trial. Colorectal Dis. 2024 Mar;26(3):545-553. doi: 10.1111/codi.16860. Epub 2024 Jan 15. PMID 38225857
- [Derived] Molenaar CJ, van Rooijen SJ, Fokkenrood HJ, Roumen RM, Janssen L, Slooter GD. Prehabilitation versus no prehabilitation to improve functional capacity, reduce postoperative complications and improve quality of life in colorectal cancer surgery. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013259. doi: 10.1002/14651858.CD013259.pub3. PMID 37162250
- [Derived] Molenaar CJ, van Rooijen SJ, Fokkenrood HJ, Roumen RM, Janssen L, Slooter GD. Prehabilitation versus no prehabilitation to improve functional capacity, reduce postoperative complications and improve quality of life in colorectal cancer surgery. Cochrane Database Syst Rev. 2022 May 19;5(5):CD013259. doi: 10.1002/14651858.CD013259.pub2. PMID 35588252
- [Derived] Onerup A, Thorn SE, Angenete E, Bock D, Gryback Gillheimer E, Haglind E, Nilsson H. Effects of a home-based exercise program on the insulin-like growth factor axis in patients operated for colorectal cancer in Sweden: Results from the randomised controlled trial PHYSSURG-C. Growth Horm IGF Res. 2020 Apr;51:27-33. doi: 10.1016/j.ghir.2020.01.005. Epub 2020 Jan 28. PMID 32007834
- [Derived] Onerup A, Angenete E, Bock D, Borjesson M, Fagevik Olsen M, Gryback Gillheimer E, Skullman S, Thorn SE, Haglind E, Nilsson H. The effect of pre- and post-operative physical activity on recovery after colorectal cancer surgery (PHYSSURG-C): study protocol for a randomised controlled trial. Trials. 2017 May 8;18(1):212. doi: 10.1186/s13063-017-1949-9. PMID 28482864